CLINICAL TRIAL: NCT01869595
Title: Prospective Study of Study to Evaluate the Feasibility of Universal HIV Testing and Antiretroviral Treatment Regardless of CD4 Count Using the Test and Treat Strategy Among Men Who Have Sex With Men and Transgender Women in Thailand
Brief Title: Thai MSM/TG Test and Treat Study
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: National Research Council of Thailand (Other Government); Ministry of Health, Thailand (Other Government); The Government Pharmaceutical Organization (Other Government); National Health Security Office, Thailand (Other)
Responsible Party: Sponsor
Other Study IDs: MSM/TG Test and Treat Study
Record Dates: First submitted 2013-06-01; First posted 2013-06-05 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2021-07

CONDITIONS: HIV Testing Rate; Acceptance of Immediate ART
Keywords: 2000 MSM and TG sites in Bangkok,Lampang,Ubonratchathani

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objectives

1. To determine the uptake of universal HIV testing among Thai men who have sex with men (MSM) and transgender women (TG)
2. To determine the uptake of antiretroviral treatment (ART) regardless of CD4 count among Thai MSM/TG who test positive for HIV

Subject population:. Men or transgender women who have sex with men,Thai nationals, age ≥18 years old, Have engaged in anal intercourse with a man without using a condom at least one time in the last 6 months or have had at least 3 male sex partners in the last 6 months,Not known to be HIV-positive (either have never been tested for HIV or have had a previous negative HIV test)

Number of participants:2000 Thai MSM and TG with approximately 76%-90% in Bangkok, 5%-12% in Lampang and 5-12% in Ubonratchathani.

DETAILED DESCRIPTION:
All participants will receive HIV testing at baseline. The frequency of study visits to determine HIV status in HIV-negative participants will be every 6 months for a total follow up time of 24 months. Once HIV-positive status is confirmed, participants will be offered ART immediately regardless of CD4 count. Those who accept ART will be seen more frequently following ART initiation, at 2 weeks, 4 weeks, 2 months, 3 months and every 3 months thereafter until completion of 24 months of follow-up. Those who deny immediate ART will have clinic visits every 6 months to monitor HIV disease. HIV-negative participants will be asked to come for HIV re-testing every 6 months or sooner if they feel exposed to risk

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationals
2. Age >18 years
3. Men or transgender women who have sex with men
4. Have engaged in anal intercourse with a man without using a condom at least one time in the last 6 months or have had at least 3 male sex partners in the last 6 months
5. Not known to be HIV-positive (either have never been tested for HIV or have had a previous negative HIV test)
6. Have signed the consent form

Exclusion Criteria:

1. Known HIV-positive serostatus

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: men who have sex with men and transgender women in Thailand
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-11; Primary Completion 2019-12 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Primary endpoints | December 1, 2015
  * Proportion of MSM who present for testing who have not previously had an HIV test
  * Proportion of HIV-negative participants who have HIV re-testing over the study period
  * Proportion of HIV-positive participants who accept ART regardless of CD4 count

CONTACTS AND LOCATIONS:
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathum Wan, Bangkok, Thailand